CLINICAL TRIAL: NCT06435793
Title: Determining Factors of the Maximal Expiratory Pressure in Healthy Individuals: Influence of the Mouthpiece Configuration
Brief Title: Expiratory Pressure in Healthy Individuals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratory of Movement, Condorcet, Tournai, Belgium (Other)
Collaborators: University of Mons (Other)
Responsible Party: Principal Investigator, Dr F Duprez, Physiotherapist / Professor at Provincial High School Condorcet (PhD), University of Mons
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P2024/081
Record Dates: First submitted 2024-05-26; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Physiology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy subjects (Experimental)
  Interventions: Procedure: MEP measurement - Surface EMG - IOPI

INTERVENTIONS:
Procedure: MEP measurement - Surface EMG - IOPI — Participants will undergo serial expiratory maneuvers using variously-sized circular mouthpieces and a reference ovoid-shaped mouthpiece.
  At each maneuver, the maximal expiratory mouth pressure at total lung capacity will be measured, alongside with the degree of neuromuscular activation of the internal oblique and transverse abdominal muscles using surface electromyography.
  The Orbicularis Oris strength will also be measured using the Iowa Oral Performance Instrument.

SUMMARY:
The present study aims at enhancing our understanding of the influence of the mouthpiece configuration on the amplitude of oral pressures generated during a maximum expiratory pressure maneuver and on the neuromuscular recruitment of expiratory muscles (more specifically of the internal oblique and the transverse abdominal muscles).

Incidentally, it also aims at clarifying the role of orofacial muscles, if any, in the neuromuscular recruitment of the aforementioned muscles.

DETAILED DESCRIPTION:
Enhancing our understanding of the influence of the mouthpiece configuration on oral pressures and on the neuromuscular recruitment of the internal oblique and the transverse abdominal muscles during a maximum expiratory pressure (MEP) maneuver is the primary goal of this study

Maximal Respiratory Mouth Pressures (MIP and MEP):

Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) are commonly used indices to assess respiratory muscle strength at the mouth.

MIP measures the strength of inspiratory muscles, while MEP assesses expiratory muscle strength.

These measurements are simple, convenient, and noninvasive. However, clear standards for these measurements are not well-established.

Choice of Mouthpiece:

We propose exploring different mouthpiece designs to know their impact on pressure measurements.

Influence of Mouthpiece Design:

The type of mouthpiece used can affect pressure measurements. Some investigators recommend including a small leak in the measuring circuit to dissipate pressure generated in the mouth and minimize measurement errors.

However, specific studies focusing on the influence of mouthpiece design on MEP and neuromuscular recruitment of expiratory muscles (such as the internal oblique and transverse muscles) during MEP maneuvers would be valuable.

Additional Considerations:

Factors like body position (sitting vs. half-lying) may also impact pressure measurements, although no significant differences were found in one study.

Among the objectives of our study, we aim at exploring ways to improve the accuracy and reliability of respiratory pressure measurements.

In summary, understanding the impact of mouthpiece design on oral pressures during MEP maneuvers is essential for accurate assessment of respiratory muscle function. Further research in this area could provide valuable insights for clinical practice and pulmonary function laboratories.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18

Exclusion Criteria:

* Any neuromuscular disease or condition susceptible to interfere with the results
* Pregnant women
* Any contraindications to the realization of maximal expiratory maneuvers, as defined in the ATS Pulmonary Function Laboratory Management And Procedure Manual (3rd Edition)
* Excessive abdominal gird, compromising ultrasonographic positioning of electrodes or altering signal quality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-18 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-09-18 (Estimated)

PRIMARY OUTCOMES:
Maximal expiratory pressure | 120 minutes
Root mean square of the EMG signal | 120 minutes

SECONDARY OUTCOMES:
Orbicularis Oris Performance Index | 5 minutes
  Obtained after computational processing of participant photographs using a MatLab based software. This index is a newly developed marker of the Orbicularis Oris function based on different anthropometric variables
Orbicularis Oris strength | 10 minutes
  Obtained through the Iowa Oral Performance Instrument

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Legrand (MD, PhD), Principal Investigator — University of Mons; Frederic Duprez (PhD), Principal Investigator — Provincial High School of Hainaut, Condorcet; Eliot Rudy Mbolo Ebubu (MD, PhD candidate), Principal Investigator — University of Mons